CLINICAL TRIAL: NCT00446966
Title: Fish Oil to Inhibit Supraventricular Arrhythmias After Cardiac Surgery: The Fish Trial
Brief Title: Fish Oil for Reduction of Atrial Fibrillation After Cardiac Surgery
Acronym: FISH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chirag Sandesara (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Chirag Sandesara, MD, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1733860001
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; coronary artery disease bypass graft surgery
MeSH Terms: conditions — Atrial Fibrillation | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fish oil , corn oil (Experimental): Highly purified pharmaceutical grade omega three polyunsaturated fatty acids
  Interventions: Drug: Omega Three Polyunsaturated fatty acids
- placebo (Placebo Comparator): olive oil
  Interventions: Drug: Omega Three Polyunsaturated fatty acids

INTERVENTIONS:
Drug: Omega Three Polyunsaturated fatty acids — 2 grams orally twice daily pre-operatively and 2 grams orally daily after until primary endpoint or 14 days.
  Other Names: Lovaza, Omega three polyunsaturate ethyl esters

SUMMARY:
The primary objective of this study is to determine if omega-3 polyunsaturated fatty acids reduce atrial fibrillation and other outcomes after cardiac surgery. In this placebo-controlled trial, patients undergoing elective coronary artery bypass graft surgery with or without valve repair will be treated with omega-3 polyunsaturated fatty acids perioperatively. The following hypotheses will be tested: 1. omega-3 polyunsaturated fatty acids reduces the incidence of atrial fibrillation (AF) after cardiac surgery, 2. omega-3 polyunsaturated fatty acids, administered in the perioperative period for cardiac surgery, decreases postoperative complication rates, and 3. omega-3 polyunsaturated fatty acids decrease intensive care unit and hospital length-of-stay.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common complication after bypass surgery. It is a significant burden to the healthcare system because it is associated with increased hospital costs and a longer hospital length-of-stay. Atrial fibrillation occurring after bypass surgery is associated with increased morbidity and mortality. Atrial fibrillation is also associated with an increased risk for strokes, use of potentially harmful drugs, and the need for pacemaker therapy.

This study is for patients who are undergoing elective bypass surgery. Patients who meet study criteria and who consent to participate in the study will be randomized to treatment with omega-3 fatty acids or matching corn oil placebo, prior to surgery. After surgery, treatment will continue until the primary endpoint, atrial fibrillation, is reached, or 14 days, whichever is first.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years old.
* Elective coronary artery bypass (CABG) operation with or without concomitant valve surgery planned for at least 2 days after enrollment.
* Signed, documented informed consent prior to admission to the study.

Exclusion Criteria:

* Urgent or emergent bypass required to be performed <24 hrs after screening.
* Unstable angina, requiring intervention or CABG <24 hrs after screening.
* Decompensated congestive heart failure.
* Chronic, persistent atrial fibrillation - patient in atrial fibrillation at the time of screening or enrollment or scheduled for a maze procedure or pulmonary vein isolation at the time of surgery.
* Known sensitivity to Omacor (0mega-3 acid ethyl esters) and hypersensitivity to fish, fish products or corn oil.
* Patients requiring warfarin or Lovenox the 2 days prior to bypass surgery.
* Patients on Class I or III antiarrhythmic agents (quinidine, procainamide, disopyramide, flecainide, propafenone, moricizine, dofetilide, sotalol, amiodarone) or who have taken these drugs within 5 elimination half-lives of the drug (or within 2 months for amiodarone).
* Patients who are pregnant or nursing.
* Patients unable to provide/sign informed consent.
* Patients currently enrolled in another clinical trial without a 30 day washout period.
* Patients currently taking marine based omega-three fish oil supplements.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chirag M Sandesara, MD, Study Chair — Virginia Cardiovascular Associates
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandesara CM, Chung MK, Van Wagoner DR, Barringer TA, Allen K, Ismail HM, Zimmerman B, Olshansky B. A Randomized, Placebo-Controlled Trial of Omega-3 Fatty Acids for Inhibition of Supraventricular Arrhythmias After Cardiac Surgery: The FISH Trial. J Am Heart Assoc. 2012 Jun;1(3):e000547. doi: 10.1161/JAHA.111.000547. Epub 2012 Jun 22. PMID 23130134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from February 2007 to December 2009. Patients were recruited from cardiothoracic clinic.
Groups:
- Fish Oil: Highly purified pharmaceutical grade omega three polyunsaturated fatty acids
Period: Overall Study
Arm/Group | Fish Oil | Corn Oil
Started | 130 | 130
Completed | 120 | 123
Not Completed | 10 | 7
Not completed — Lost to Follow-up | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Corn Oil: Standard grade corn oil
- Total: Total of all reporting groups
Arm/Group | Fish Oil | Corn Oil | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.5) | 62 (11.4) | 62 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 28 | 64
  Male | 94 | 102 | 196
Region of Enrollment [Number; unit: participants]
  United States | 130 | 130 | 260

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Postoperative Atrial Fibrillation
Description: The primary outcome in this study is post-bypass atrial fibrillation documented by ECG or rhythm strip and requiring treatment.
Time Frame: 14 days
Population: Intention to treat
Measure: Number; unit: participants
Groups:
- Corn Oil: Corn oil
Arm/Group | Corn Oil | Fish Oil
Number analyzed (Participants) | 130 | 130
participants | 33 | 30
Statistical Analysis 1: Comparison: Corn Oil vs Fish Oil; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Corn Oil: Standard corn oil
Arm/Group | Fish Oil | Corn Oil
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/130
Other Adverse Events (participants affected / at risk) | 0/130 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No